CLINICAL TRIAL: NCT04037423
Title: European Database on Catheter-directed Treatment of Pulmonary Embolism.
Acronym: EuroPE-CDT
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: EuroPE-CDT
Record Dates: First submitted 2019-07-22; First posted 2019-07-30 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Acute Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PE patients treated with CDT: Acute pulmonary embolism patients undergoing catheter-directed embolectomy.

SUMMARY:
The main goals of EuroPE-CDT is to assess the currently applied catheter-directed treatment (CTD) techniques and strategies in pulmonary embolism (PE) patients and to determine the short term efficacy and safety of this invasive procedure.

DETAILED DESCRIPTION:
This is a prospective (and retrospective, if required data are available), non-interventional, multicenter study. We intend to obtain data on basic patients characteristics, pulmonary embolism severity, catheter-directed treatment procedures and short term outcome. We are planning to include approximately 150-200 patients suitable for analysis by the end of 2020. Anonymized data of consecutive PE patients treated with CTD in European centers will be collected in the database.

ELIGIBILITY:
Inclusion Criteria:

* acute pulmonary embolism
* catheter-directed embolectomy

Exclusion Criteria:

* appropriate data not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Survival | 30 days after the procedure
  Short-time follow-up

SECONDARY OUTCOMES:
Complications | During hospitalisation (estimated 10 days)
  Any procedure-related complications, such as:
  * local hematoma,
  * hemoptysis,
  * pulmonary artery injury,
  * contrast-induced nephropathy,
  * renal replacement therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Purszczyk, prof., Study Chair — Medical University of Warsaw
Locations (1):
- Department of Internal Medicine & Cardiology with the Centre for Management of Venous Thromboembolic Disease, Medical University of Warsaw, Warsaw, Poland